CLINICAL TRIAL: NCT04560114
Title: Effect of Inhaled Aromatherapy on Chemo-Induced Nausea Vomiting (NCVI): CINVAROM (Chemotherapy Induced Nausea Vomiting and AROMatherapy)
Acronym: CINVAROM
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Centre Francois Baclesse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CINVAROM
Record Dates: First submitted 2020-09-17; First posted 2020-09-23 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Nausea and Vomiting; Aromatherapy; Essential Oil; Suportive Care
MeSH Terms: conditions — Nausea; Vomiting | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Open, prospective, single-center phase 2 study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Essential oils (Experimental): Inhalation will be carried out via an inhaler stick containing essential oils (Mentha x Piperita; Citrus Limon; Zingiber Officinale)
  Interventions: Drug: Essential oils

INTERVENTIONS:
Drug: Essential oils — The patient will be invited to inhale the essential oils via the stick:
  * 4 times a day before each meal and snack.
  * if necessary when nausea appears, as many times as he deems necessary.

SUMMARY:
The investigator wish to provide a blend of two essential oils with comparable antiemetic properties; Peppermint essential oil (Mentha x Piperita) and lemon tree essential oil (Citrus Limon). Dry inhalation of these essential oils is safe, but effectiveness has not been determined. Studies on the subject present a questionable methodology. This is why we are proposing this study to measure the effectiveness of this mixture of essential oils on chemo-induced nausea and vomiting.

This study is a first step before a possible study to compare the effects of essential oils with those of a placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients will be eligible if:

* Aged over 18,
* Presenting a solid tumor in the 1st line of chemotherapy administered by intravenous route;
* Treated with adjuvant or neoadjuvant chemotherapy;
* Affiliated with a social security scheme;
* Able to understand the meaning of the questions asked;
* Having given their written consent to participate in the study;
* Whether or not treated with surgery and radiotherapy before entering the study

Exclusion Criteria:

Patients who:

* Do not give their consent to participate;
* Do not master the French language;
* Are deprived of their liberty, under guardianship or curatorship;
* Suffer from cognitive deficits or associated psychiatric disorders that could compromise their ability to participate in the study (eg: schizophrenia);
* Are undergoing radiotherapy;
* Must receive a combination of radio-chemotherapy;
* Whose chemotherapy protocol is composed of several chemotherapy administrations per week during a course of treatment;
* have been previously treated with chemotherapy;
* Have an occlusive syndrome;
* Have primary cancer of the central nervous system or brain metastases;
* Have cancer of the Upper Aero Digestive Tract;
* Simultaneously participate in a therapeutic clinical trial;
* Have an intolerance to a component of essential oils;
* Pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2020-12-14 (Actual); Primary Completion 2021-09-21 (Actual); Study Completion 2023-06-30 (Actual)

PRIMARY OUTCOMES:
Number of episodes of nausea and vomiting | 4 days after the first cycle of chemotherapy

SECONDARY OUTCOMES:
Number of episodes of nausea and vomiting | 4 days after the third cycle
Anxiety with self-questionnaire HADS | 21 days after the third cycle

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Francois Baclesse, Caen, France

IPD SHARING:
Plan to Share IPD: Undecided